CLINICAL TRIAL: NCT02355470
Title: GIFTSS (Giving Information for Trauma Support and Safety): A College Health Center-based Alcohol and Sexual Violence Intervention
Brief Title: College Health Center-based Alcohol and Sexual Violence Intervention
Acronym: GIFTSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Elizabeth Miller, Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14110392
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Sexual Assault; Alcohol Consumption; Intimate Partner Violence
Keywords: Sexual assault; Alcohol consumption; Intimate partner violence
MeSH Terms: conditions — Alcohol Drinking | interventions — Safety; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Participants will receive the GIFTSS intervention provided by college health center staff and clinicians
  Interventions: Behavioral: GIFTSS
- Control (Active Comparator): Participants will receive a brief alcohol use reduction intervention based on NIAAA guidelines provided by college health center staff and clinicians
  Interventions: Behavioral: Brief alcohol use intervention

INTERVENTIONS:
Behavioral: GIFTSS — Universal education and brief counseling regarding sexual violence
  Other Names: Giving Information for Trauma Support and Safety
  Arms: Intervention
Behavioral: Brief alcohol use intervention — Brief education and counseling intervention to promote safer alcohol use, reduce binge drinking
  Arms: Control

SUMMARY:
This study will offer the first formal assessment for sexual violence (SV) in the college student health center setting, developed for a high risk group of college students, and is designed to facilitate patient and provider comfort in discussing sexual violence and related abusive experiences (including the role of alcohol) via semi-scripted screening tools. The intervention specifically involves the training of all clinical staff (health educators, counselors, medical assistants, nurses, and clinicians) to deliver a universal education and brief counseling intervention titled GIFTSS (Giving Information for Trauma Support and Safety) to all clients seeking college health services integrated into usual clinical practice, provide universal education about SV regardless of disclosure, counsel clients on harm reduction strategies to reduce risk for SV, and provide supported referrals to sexual assault advocates, with the goal of reducing SV among college students.

DETAILED DESCRIPTION:
This is a stakeholder-engaged longitudinal study to test, via a 2-armed cluster randomized controlled trial , a brief harm reduction intervention to reduce risk for sexual violence among male and female college students ages 18-24 receiving care from college student health services (K = 28 colleges; baseline N = 2295). Sexual violence (SV) (including sexual coercion, non-consensual sexual contact, and rape) is common among college women, and over three quarters of women who have been sexually assaulted report that the first of such experiences occurred before the age of 25. Alcohol-related SV, in particular, is highly prevalent on college campuses, with about half of sexual assault cases occurring in the context of victim and/or perpetrator intoxication. Multiple pathways have been implicated in this association between alcohol and SV, with social norms regarding alcohol consumption and expectations for SV facilitating both the occurrence and underreporting of such violence. College student health centers remain an untapped setting to reach youth for both SV prevention and intervention. This study draws on several intervention studies by the investigative team, integrating successful components from each: 1) the bystander approach in which individuals are taught skills as active interveners in SV prevention rather than responding with apathy or tolerance is an effective strategy for promoting change within social contexts; 2) universal education about SV regardless of disclosure in the clinical setting can result in increased recognition of SV and use of relevant services; and 3) harm reduction strategies introduced by clinicians can increase intentions to use strategies to help oneself and friends that increase safety. The brief counseling intervention uses a palm-size educational card with information about SV and harm reduction given to all patients during clinical encounters. GIFTSS (Giving Information for Trauma Support and Safety) provides (a) patient education and assessment regarding SV; (b) discussion of harm reduction behaviors to reduce risk of SV for self and peers (including bystander intervention); and (c) supported referrals to victim services. Interventions effective in reaching more college-age young adults who either witness or experience SV are needed. College student health centers randomized into the GIFTSS intervention arm will receive training in this brief intervention integrated into routine college health visits. The control sites will receive a brief alcohol intervention. Compared to controls, male and female clients receiving the GIFTSS intervention are expected to have greater recognition of what constitutes SV and alcohol-related sexual risk (primary outcome), recognition of sexual coercion, self-efficacy to obtain sexual consent, self-efficacy to enact harm reduction strategies, intentions to intervene, and knowledge of and self-efficacy to use SV-related services (Aim 1). Among participants who have witnessed peer SV, those receiving GIFTSS will be more likely to report interventions to interrupt peer's harmful behaviors (Aim 2). Clients with SV victimization history who receive GIFTSS are expected to be more likely to disclose SV during their clinic visit, report greater use of SV-related services, and report less recent SV victimization at follow up compared to control clients (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-24
* Able to read English
* Seeking care at the college health center for any reason

Exclusion Criteria:

* Younger than 18 or older than 24 years
* Not seeking care at the college health center

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2295 (Actual)
Dates: Start 2015-08; Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Change in recognition of alcohol-related sexual violence and sexual risk from baseline to follow up | 4 months and 12 months
  Changes in overall mean knowledge score measuring recognition of what constitutes sexual violence and the role of alcohol in risk for sexual violence comparing baseline and follow up

SECONDARY OUTCOMES:
Change in self-efficacy to use harm reduction strategies | 4 months and 12 months
  Post-intervention levels of self-efficacy to use specified harm reduction strategies to reduce risk for sexual violence adjusting for baseline general self-efficacy
Change in knowledge of sexual violence related services from baseline to follow up | 4 months and 12 months
  Knowing about specified sexual violence related services comparing baseline and follow up summary scores
Change in self-efficacy to use sexual violence related services | 4 months and 12 months
  Changes in mean score measuring self-efficacy to use violence related services comparing baseline and follow up
Change in intentions to intervene from baseline to follow up | 4 months and 12 months
  Proclivity to intervene when witnessing disrespectful and harmful behaviors among peers comparing baseline and follow up mean scores on a scale assessing likelihood of trying to stop harmful behaviors among peers
Change in positive bystander behaviors from baseline to follow up | 4 months and 12 months
  Assessment of recent positive bystander behavior in students when witnessing disrespectful and harmful behaviors among peers comparing baseline and follow up summary scores. Students report if they have witnessed peers' abusive behaviors in recent months and if witnessed, how they responded (whether they intervened to interrupt the behavior)
Change in recognition of sexual coercion from baseline to follow up | 4 months and 12 months
  Changes in mean score measuring recognition of what constitutes sexual coercion comparing baseline and follow up
Change in self-efficacy to obtain sexual consent | 4 months and 12 months
  Changes in mean score assessing self-efficacy to obtain sexual consent comparing baseline and follow up

OTHER OUTCOMES:
Change in sexual violence victimization from baseline to follow up | 4 months and 12 months
  Among those reporting exposure to sexual violence at baseline, summary score of any sexual violence victimization (including partner violence, forced alcohol consumption prior to sex, respondent alcohol consumption prior to sex, unwanted sexual experiences), comparing the time before the intervention to after the intervention
Sexual violence disclosure to health center provider | At time of baseline clinical encounter, 4 months, and 12 months
  Among those reporting exposure to sexual violence, disclosed to health center provider during health center visits
Change in use of sexual violence related services | 12 months
  Any use of sexual violence related services (summary score)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Coulter RWS, Gartner RE, Cramer C, Smith EK, Abebe KZ, Miller E. Universal Sexual Violence Intervention Effects in a Cluster-Randomized Trial: Moderation by Sexual Orientation. J Interpers Violence. 2025 Feb;40(3-4):582-606. doi: 10.1177/08862605241253031. Epub 2024 May 18. PMID 38761368
- [Derived] Anderson JC, Peruggia G, Miller-Walfish S, Talis J, Burrell C, Hayes M, Miller E. A case series measuring campus and clinic level factors during implementation of a sexual violence prevention intervention in campus health and counseling centers: does environment matter? Implement Sci Commun. 2023 Jul 31;4(1):88. doi: 10.1186/s43058-023-00467-7. PMID 37525258
- [Derived] Miller E, Jones KA, McCauley HL, Rofey DL, Clark DB, Talis JM, Anderson JC, Chugani CD, Coulter RWS, Abebe KZ. Cluster Randomized Trial of a College Health Center Sexual Violence Intervention. Am J Prev Med. 2020 Jul;59(1):98-108. doi: 10.1016/j.amepre.2020.02.007. Epub 2020 Apr 30. PMID 32362510
- [Derived] Abebe KZ, Jones KA, Rofey D, McCauley HL, Clark DB, Dick R, Gmelin T, Talis J, Anderson J, Chugani C, Algarroba G, Antonio A, Bee C, Edwards C, Lethihet N, Macak J, Paley J, Torres I, Van Dusen C, Miller E. A cluster-randomized trial of a college health center-based alcohol and sexual violence intervention (GIFTSS): Design, rationale, and baseline sample. Contemp Clin Trials. 2018 Feb;65:130-143. doi: 10.1016/j.cct.2017.12.008. Epub 2017 Dec 26. PMID 29287667